CLINICAL TRIAL: NCT03707015
Title: Internal Limiting Membrane Flap in the Management of Retinal Detachment Due to Paracentral Retinal Breaks
Status: Completed | Type: Observational
Sponsor: San Ni Chen (Other)
Responsible Party: Sponsor-Investigator, San Ni Chen, Department of Ophthalmology, Changhua Christian Hospital
Organization: Changhua Christian Hospital (Other)
Other Study IDs: 180315
Record Dates: First submitted 2018-10-08; First posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Retinal Detachment; Surgery
Keywords: Retinal Detachment; internal limiting membrane flap; retinal paracentral breaks
MeSH Terms: conditions — Retinal Detachment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To describe the technique and outcomes of using either inverted or free internal limiting membrane flap in the management of retinal detachment due to paracentral retinal breaks.

DETAILED DESCRIPTION:
This retrospective observational case series includes nine patients received surgery for retinal detachment due to paracentral retinal breaks developed either from primary rhegmatogenous orgin, or secondary iatrogenic retinal breaks after prior membrane peeling or during surgery for tractional retinal detachment. Either inverted or free internal limiting membrane flaps were inserted in the identified breaks, followed by air fluid exchange and gas tamponade. Visual acuity and structural changes were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with retinal detachment and posterior paracentral retinal breaks located within the equator from January 2017 to January 2018

Exclusion Criteria:

* Patient with macular hole
* Patient with other ocular diseases including ocular hypertension, optic nerve atrophy, glaucoma or chronic uveitis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We included patients with retinal detachment and posterior paracentral retinal breaks located within the equator from January 2017 to January 2018. Eyes with macular hole were excluded. All of the cases underwent standard pars plana vitrectomy using the ILM flap technique, accompanied by extended gas tamponade without laser retinopexy
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
re-attachment rate of retinal detachment | within 3 months postoperatively
  re-attachment of retina through examination including fundoscopic exam and optical coherent tomography exam

SECONDARY OUTCOMES:
visual acuity | within 3 months postoperatively
  visual acuity in logMAR

CONTACTS AND LOCATIONS:
Overall Officials: San-Ni Chen, M.D, Principal Investigator — Changhua Christian Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Chen SN, Yang CM. Inverted Internal Limiting Membrane Insertion for Macular Hole-Associated Retinal Detachment in High Myopia. Am J Ophthalmol. 2016 Feb;162:99-106.e1. doi: 10.1016/j.ajo.2015.11.013. Epub 2015 Nov 12. PMID 26582311
- [Result] Chen SN, Hsieh YT, Yang CM. Multiple Free Internal Limiting Membrane Flap Insertion in the Treatment of Macular Hole-Associated Retinal Detachment in High Myopia. Ophthalmologica. 2018;240(3):143-149. doi: 10.1159/000487337. Epub 2018 Jun 6. PMID 29874671
- [Derived] Chen YC, Yang CM, Chen SN. Internal Limiting Membrane Flap in the Management of Retinal Detachment due to Paracentral Retinal Breaks. J Ophthalmol. 2019 Jan 21;2019:4303056. doi: 10.1155/2019/4303056. eCollection 2019. PMID 30805208